CLINICAL TRIAL: NCT03823235
Title: Humidified Incubator Effect on Live Birth Rate After ICSI
Brief Title: Humidified Culture and Live Birth After ICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibn Sina Hospital (Other Government)
Collaborators: Banoon IVF Center (Other); Quena IVF Center (Unknown); Amshag IVF Center (Unknown)
Responsible Party: Principal Investigator, Muhammad Fawzy, Lab Director, Ibn Sina Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IbnSina-Humidity
Record Dates: First submitted 2019-01-27; First posted 2019-01-30 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culture of human embryo in non-humidified incubator (Experimental): Embryo culture after in vitro fertilization in incubator with no humidity
  Interventions: Other: Human embryo culture
- Culture of human embryo in humidified incubator (No Intervention): Embryo culture after in vitro fertilization in incubator with humidity

INTERVENTIONS:
Other: Human embryo culture — humidifed or dry incubator
  Arms: Culture of human embryo in non-humidified incubator

SUMMARY:
Humidity for human embryo culture has been raised as essential with advantageous effect on clinical pregnancy and ongoing pregnancy after ICSI compared with a dry incubator. Whether the deleterious effect of dry culture would have an extended effect reaches the live birth rate needs to be examined. This RCT is to examine the effect of dry and humidified culture on live birth rates after ICSI.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing a first or second ICSI attempts
* Primary or secondary infertility with a BMI of < 31 kg/m2
* Duration of infertility of ≥ 18 months and normal baseline ultrasonography
* 18 to 40 years of age
* Tubal factor, male factor, polycystic ovary, unexplained infertility or combined factors
* Tubal factors

Exclusion Criteria:

* Surgically-retrieved, frozen-thawed and pinpoint sperm or globozoospermia
* Thin endometrium
* Uterine anomaly and adhesion
* Adenomyosis
* Submucous myoma
* Endometriosis
* Severe medical condition

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1837 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Live birth rate | 30 weeks
  Viable neonate after 30 weeks of gestation per initiated cycle

SECONDARY OUTCOMES:
Cumulative live birth rate | One year
  Viable neonate after 30 weeks of gestation after one fresh and/or one frozen-warmed transfer per initiated cycle
Ongoing pregnancy rate | 12 weeks of gestation
  Continued pregnancy after 12 weeks of gestation per initiated cycle
Cumulative ongoing pregnancy rate | 12 weeks of gestation
  Continued pregnancy after 12 weeks of gestation per initiated cycle within one year of randomization
Clinical pregnancy rate | 7 weeks of gestation
  Ultrasound detect heartbeat after 7 weeks of gestation per initiated cycle
Cumulative clinical pregnancy rate | 7 weeks of gestation
  Ultrasound detect heartbeat after 7 weeks of gestation per initiated cycle within one year of randomization
Implantation rate | 7 weeks of gestation
  Number of sacs with a heartbeat per number of embryo transferred
Cumulative implantation rate | 7 weeks of gestation
  Number of sacs with a heartbeat per number of embryo transferred within one year of randomization
Ongoing implantation rate | 12 weeks of gestation
  Number of sacs with a heartbeat per number of embryo transferred
Cumulative ongoing implantation rate | 12 weeks of gestation
  Number of sacs with a heartbeat per number of embryo transferred within one year of randomization
Preterm birth rate | 37 weeks
  number of babies born before 37 weeks of gestation per total birth
Very preterm birth | 32 weeks
  number of babies born before 32 weeks of gestation per total birth
Low birth weight rate | 40 weeks of gestation
  number of babies with < 2500 gm per total birth
Fertilization rate | 6 days of culture
  fertilized oocytes with two pronuclei per Metaphase II injected
Cleavage rate | 6 days of culture
  Cleaved embryo per fertilized oocyte
Rate of high-quality day-3 embryos | 6 days of culture
  Embryos with seven or eight blastomeres of appropriate-size, and < 10% fragmentation by volume per fertilized oocyte
Blastocyst formation rate | 6 days of culture
  Formed blastocyst on day 5/6 from fertilized oocytes
Rate of high-quality blastocyst | 6 days of culture
  Blastocysts ≥ 3.1.1 grade per fertilized oocyte
Rate of utilizable blastocyst | 6 days of culture
  Transferred and cryopreserved blastocysts from fertilized oocytes

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Qena Fertility Center, Qina, Qena Governorate
  - Banon Assiut, Asyut
  - IbnSina IVF Center, Sohag

IPD SHARING:
Plan to Share IPD: No